CLINICAL TRIAL: NCT06436313
Title: The Value of Virtual Education on Deep Brain Stimulation for Surgical Candidates
Brief Title: DBS Virtual Learning Experience
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Alfonso Fasano, Professor, Department of Medicine, Division of Neurology at University of Toronto, Toronto Western Hospital, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-5018
Record Dates: First submitted 2024-05-24; First posted 2024-05-31 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational Group (Experimental): Patients will receive two extra virtual educational sessions.
  Interventions: Other: Educational Sessions
- Standard-of-Care (No Intervention): Patients will not receive any extra educational sessions. Their education will be provided as per standard-of-care by the clinical team.

INTERVENTIONS:
Other: Educational Sessions — Two online educational sessions will be organized before DBS surgery. These will be scheduled between consultation with the neurologist and the consultation with the neurosurgeon. Each virtual session will last about 1 hour. Patients can login from home, together with their caregivers. The virtual sessions will be held on MS Teams virtual platform.
  One of the sessions will include a DBS patient where patients will have the opportunity to ask peer-to-peer questions. The session includes testimonials from patient before and after their surgery.
  The second session (about two weeks later) is a summary presentation, a quiz and time for Q&A. During one of the sessions (first or second), a DBS patient (who has been implanted) can be invited to participate togive the attendees the opportunity to ask peer-to-peer questions. The quiz contains questions to assess the patients' knowledge of DBS.
  Arms: Educational Group

SUMMARY:
The success of Deep Brain Stimulation (DBS) is more correlated to fulfillment of patients' expectations, than merely improvement of motor status1. Therefore, it is of utmost importance to inform the DBS candidates as good as possible to set realistic expectations. Currently, the patient - most of the time accompanied by a family member - is informed about the surgery and its benefits and risks during the outpatient consultation of the neurologist, and later on during the consultation of the neurosurgeon. Written information is provided in the form of a booklet that the patients take home.

Due to the large amount of information, not all of it can be captured by the patient. Therefore, we would like to investigate whether an additional online immersive educational session on DBS would better educate the patient. The online session is a 1-hour video call with a small group of DBS candidates and their caregivers, lead by DBS experts, where testimonials of other patients are shown, together with multiple infographics. Two weeks later their will be a second online session summarizing the information and providing the opportunity for Q&A.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of any age over 18 who are capable of understanding and granting informed consent.
2. Consecutive enrollment of Parkinson's disease patients, eligible for DBS surgery who will be operated in Toronto Western Hospital.
3. Targets of surgery (STN or GPi) equally in each study arm.
4. Patients must be able to follow the assessment procedure.

Exclusion Criteria:

1. people with limited digital skills (to the discretion of the PI).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
The Parkinson's Disease Questionnaire (PDQ-39) | Baseline, 3 months post op
  This questionnaire assesses how often people with Parkinson's experience difficulties. across 8 dimensions of daily living. The total score for each dimension ranges from 0 (never have difficulty) to 100 (always have difficulty). Lower scores indicate better quality of life.
MDS-UPDRS (Movement Disorders Society Unified Parkinson's Disease Rating Scale) | Baseline, 3 months post op
  Is composed of 4 parts4. Part 1 in on the non-motor aspects of experiences of daily living, with the first half begin rated by the health care professional, based on input from the patient and the caregiver; and the second half a patient questionnaire. Part 2 is on the motor aspects of experiences of daily living, which is a questionnaire filled out by the patient and the caregiver. In the 3rd part the motor condition of the patient evaluated by the physician or nurse practitioner, in meds-ON and DBS-ON condition. The fourth and final part evaluates the motor complications and is rated by the health care professional, based on input from the patient and the caregiver.
  The total score on the MDS-UPDRS ranges from 0 to 260. The score indicates:
  0: No disability 260: Total disability.
Parkinson Anxiety Scale (PAS) | Baseline, 3 months post op
  is a 12-item observer or patient-rated scale with three subscales, for persistent and episodic anxiety, and avoidance behaviour. The total score on the PAS can range from 0 to 48.
  Higher scores indicate greater experiences of anxiety
The Beck Depression Inventory (BDI) | Baseline, 3 months post op
  Is a 21-items questionnaire that is filled out by the patient to self-rate mood-related statements. The total score can range from 0 to 63.
  Higher scores indicate greater severity of depressive symptoms.
Structured survey | Baseline, one day before surgery, 3 months post op
  Assesses the level of knowledge (score range: 0-110), anxiety (score range: 0-100), expectation (score range: 0-100), satisfaction (score range: 0-80).

CONTACTS AND LOCATIONS:
Locations (1):
- Movement Disorders Centre - Toronto Western Hospital, Toronto, Ontario, Canada